CLINICAL TRIAL: NCT00270998
Title: ATLAS: Ambulatory Treatments for Leakage Associated With Stress, A Randomized Trial of Pelvic Muscle Exercise Versus Incontinence Pessary Versus Both for Women With Stress or Mixed Urinary Incontinence
Brief Title: ATLAS: Ambulatory Treatments for Leakage Associated With Stress
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NICHD Pelvic Floor Disorders Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PFDN 13
Record Dates: First submitted 2005-12-27; First posted 2005-12-29 (Estimated); Results first posted 2017-08-10 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-04

CONDITIONS: Stress Urinary Incontinence; Urinary Incontinence
Keywords: Stress urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intravaginal Pessary (Experimental): Pessary restores continence by stabilization of the proximal urethra and urethrovesical junction, facilitating pressure transmission to the proximal urethra.
  Interventions: Device: Intravaginal Pessary
- Behavioral Therapy (Experimental): Pelvic floor muscle training and exercise which includes strong contraction of the pelvic floor muscles to prevent incontinence by occluding the urethra and regular practice can improve pelvic muscle support.
  Interventions: Behavioral: Behavioral Therapy
- Pessary combined with behavioral therapy (Experimental): Combination of the explanations above.
  Interventions: Device: Pessary combined with behavioral therapy

INTERVENTIONS:
Behavioral: Behavioral Therapy — Pelvic muscle training and exercises
  Arms: Behavioral Therapy
Device: Intravaginal Pessary — Intravaginal pessary
  Arms: Intravaginal Pessary
Device: Pessary combined with behavioral therapy — Intravaginal pessary and behavioral therapy
  Arms: Pessary combined with behavioral therapy

SUMMARY:
Stress urinary incontinence is the uncontrollable leakage of urine with physical effort or stress, such as coughing, sneezing, or exercise. Treatment for stress incontinence can be surgical or non-surgical. Different non-surgical treatments include pelvic muscle exercises and pessary use. Pelvic muscle exercises (often known as "Kegel" exercises) train and strengthen the pelvic muscles and improve incontinence. A pessary is a medical device that fits inside the vagina to give the urethra and bladder extra support and prevent or reduce urinary incontinence. Exercises and pessary use can help women with stress incontinence but it is not known which treatment is better, or if a combination of the two treatments at the same time is best. This study will determine whether pelvic muscle training and exercises, pessary use, or a combination of both exercises and pessary is most effective at improving incontinence in women. The study's primary hypothesis is that pessary use is more effective than pelvic muscle exercises after 3 months of treatment.

DETAILED DESCRIPTION:
Women commonly have symptoms of stress urinary incontinence (leakage with physical stress such as coughing or sneezing) and urinary urgency or urge incontinence (leakage associated with the overwhelming urge to urinate). Non-surgical treatment is usually offered as first-line therapy, such as pelvic muscle exercises ("Kegel" exercises) or pessary use. A pessary is a small ring that fits inside the vagina. Pelvic muscle training and exercises may help incontinence by increased awareness and strength of the muscles that are used in holding the urethra closed. Pessary use may help incontinence by providing more support to the bladder and urethra. Both treatments can be helpful in reducing or eliminating incontinence, but it is not known which treatment is better. The study will compare the level of improvement with pelvic muscle exercises, pessary use, and a combination of both exercises and pessary.

Women with stress or mixed urinary incontinence will be randomly assigned to 1 of 3 groups: (1) pelvic muscle training and exercises; (2) pessary use; and (3) both exercises and pessary. Women in the exercises groups will have 4 visits over 8 weeks with a specially trained therapist for pelvic muscle training and exercises. Women in the pessary group will be fitted with a pessary to be worn continuously. Assessments will include questionnaires, bladder diary, and physical examination. Follow-up evaluations occur at 3 months, 6 months (by telephone only), and 1 year after initial treatment.

Comparisons: The level of improvement after treatment will be compared in the 3 groups. In addition, women in the 3 groups will record the number of accidental leakage episodes by bladder diary; and the frequency of those episodes will be compared in the 3 groups. Other aspects of health, including health-related quality of life, will be compared in the 3 groups.

ELIGIBILITY:
Inclusion Criteria:

* Stress urinary incontinence or stress-predominant mixed urinary incontinence, with at least 2 episodes of stress incontinence on 7-day bladder diary and the number of stress incontinence episodes exceeding the number of urge incontinence episodes.
* Urinary incontinence for at least three months.
* Ambulatory adult women.
* Stage 0-I-II pelvic organ prolapse.

Exclusion Criteria:

* Continual urine leakage.
* Pregnancy or planning pregnancy within 1 year.
* Active urinary tract infection.
* Urinary retention.
* Currently on medication for incontinence.
* Currently using a pessary.
* Neurologic condition that affects bladder function.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2005-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly E Richter, PhD, MD, Study Chair — University of Alabama at Birmingham
Locations (8):
- United States (8):
  - University of Alabama, Birmingham, Alabama
  - University of California, San Diego Medical Center, La Jolla, California
  - Loyola University, Maywood, Illinois
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Texas Southwestern, Dallas, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Richter HE, Burgio KL, Goode PS, Borello-France D, Bradley CS, Brubaker L, Handa VL, Fine PM, Visco AG, Zyczynski HM, Wei JT, Weber AM; Pelvic Foor Desorders Network. Non-surgical management of stress urinary incontinence: ambulatory treatments for leakage associated with stress (ATLAS) trial. Clin Trials. 2007;4(1):92-101. doi: 10.1177/1740774506075237. PMID 17327249
- [Result] Richter HE, Burgio KL, Brubaker L, Nygaard IE, Ye W, Weidner A, Bradley CS, Handa VL, Borello-France D, Goode PS, Zyczynski H, Lukacz ES, Schaffer J, Barber M, Meikle S, Spino C; Pelvic Floor Disorders Network. Continence pessary compared with behavioral therapy or combined therapy for stress incontinence: a randomized controlled trial. Obstet Gynecol. 2010 Mar;115(3):609-617. doi: 10.1097/AOG.0b013e3181d055d4. PMID 20177294
- [Derived] Borello-France D, Burgio KL, Goode PS, Ye W, Weidner AC, Lukacz ES, Jelovsek JE, Bradley CS, Schaffer J, Hsu Y, Kenton K, Spino C; Pelvic Floor Disorders Network. Adherence to behavioral interventions for stress incontinence: rates, barriers, and predictors. Phys Ther. 2013 Jun;93(6):757-73. doi: 10.2522/ptj.20120072. Epub 2013 Feb 21. PMID 23431210
- [Derived] Schaffer J, Nager CW, Xiang F, Borello-France D, Bradley CS, Wu JM, Mueller E, Norton P, Paraiso MF, Zyczynski H, Richter HE. Predictors of success and satisfaction of nonsurgical therapy for stress urinary incontinence. Obstet Gynecol. 2012 Jul;120(1):91-7. doi: 10.1097/AOG.0b013e31825a6de7. PMID 22914396
- [Derived] Kenton K, Barber M, Wang L, Hsu Y, Rahn D, Whitcomb E, Amundsen C, Bradley CS, Zyczynski H, Richter HE; Pelvic Floor Disorders Network. Pelvic floor symptoms improve similarly after pessary and behavioral treatment for stress incontinence. Female Pelvic Med Reconstr Surg. 2012 Mar-Apr;18(2):118-21. doi: 10.1097/SPV.0b013e31824a021d. PMID 22453323
- [Derived] Barber MD, Chen Z, Lukacz E, Markland A, Wai C, Brubaker L, Nygaard I, Weidner A, Janz NK, Spino C. Further validation of the short form versions of the Pelvic Floor Distress Inventory (PFDI) and Pelvic Floor Impact Questionnaire (PFIQ). Neurourol Urodyn. 2011 Apr;30(4):541-6. doi: 10.1002/nau.20934. Epub 2011 Feb 22. PMID 21344495
- [Derived] Barber MD, Spino C, Janz NK, Brubaker L, Nygaard I, Nager CW, Wheeler TL; Pelvic Floor Disorders Network. The minimum important differences for the urinary scales of the Pelvic Floor Distress Inventory and Pelvic Floor Impact Questionnaire. Am J Obstet Gynecol. 2009 May;200(5):580.e1-7. doi: 10.1016/j.ajog.2009.02.007. PMID 19375574
- See also: Website of the National Institute of Child Health and Human Development, which funds the Pelvic Floor Disorders Network — http://www.nichd.nih.gov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 740 women were screened for symptoms of stress only or mixed incontinence symptoms and age of at least 18 years old. 294 did not meet inclusion criteria, one refused to participate and 445 were enrolled.
Groups:
- Pessary: Intravaginal incontinence pessary
- Combination of Pessary and Behavioral Therapy: Treatment is a combination of both pessary and pelvic muscle exercises
Period: 3 Month Follow-up
Arm/Group | Pessary | Behavioral Therapy | Combination of Pessary and Behavioral Therapy
Started | 149 | 146 | 150 (1 participant randomized to combined found ineligible at first treatment visit, removed from study.)
Completed | 110 | 124 | 132
Not Completed | 39 | 22 | 18
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 2 | 1
Not completed — Withdrawal by Subject | 11 | 14 | 15
Not completed — Pessary did not fit | 12 | 0 | 0
Not completed — Personal/family health | 1 | 1 | 0
Not completed — Received/desired alternate treatment | 13 | 5 | 2
Period: 12 Month Follow-up
Arm/Group | Pessary | Behavioral Therapy | Combination of Pessary and Behavioral Therapy
Started | 110 | 124 | 132
Completed | 96 | 99 | 111
Not Completed | 14 | 25 | 21
Not completed — Lack of Efficacy | 5 | 4 | 3
Not completed — Withdrawal by Subject | 7 | 12 | 16
Not completed — Pessary did not fit | 1 | 0 | 0
Not completed — Personal/family health | 0 | 5 | 1
Not completed — Received/desired alternate treatment | 1 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Pessary: Intravaginal pessary
- Combination of Pessary and Behavioral Therapy: Treatment includes a combination of both pessary and pelvic muscle exercises
- Total: Total of all reporting groups
Arm/Group | Pessary | Behavioral Therapy | Combination of Pessary and Behavioral Therapy | Total
Number analyzed (Participants) | 149 | 146 | 150 | 445
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (11.0) | 49.6 (13.0) | 49.5 (11.8) | 49.8 (11.9)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 149 | 146 | 150 | 445
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 126 | 132 | 122 | 380
  Black or African American | 15 | 10 | 20 | 45
  Other | 8 | 4 | 8 | 20
Vaginal Deliveries [Median (Inter-Quartile Range); unit: deliveries] | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]
Menstrual Status [Count of Participants; unit: Participants]
  Pre-menopausal | 75 | 71 | 68 | 214
  Post-menopausal | 60 | 62 | 66 | 188
  Not sure | 14 | 13 | 16 | 43
Prior Nonsurgical UI [Count of Participants; unit: Participants] | 30 | 35 | 27 | 92
Prior UI Surgery [Count of Participants; unit: Participants] | 10 | 7 | 10 | 27
Hysterectomy [Count of Participants; unit: Participants] | 39 | 39 | 32 | 110
Incontinence Type [Count of Participants; unit: Participants]
  Stress Only | 69 | 65 | 70 | 204
  Mixed | 80 | 81 | 80 | 241
Incontinence Frequency [Count of Participants; unit: Participants]
  14 or more episodes per wk | 68 | 67 | 67 | 202
  Fewer than 14 episodes per wk | 81 | 79 | 83 | 243
Currently Receiving Estrogen Therapy [Count of Participants; unit: Participants] | 27 | 24 | 16 | 67

OUTCOME MEASURES:

1. Primary Outcome: "Much Better" or "Very Much Better" on PGI-I at 3 Months
Description: PGI-I, Patient Global Impression of Improvement, is a five-point scale that ranges from "not at all" to "very much better." Participants were considered a success if they responded "much better" or "very much better," or a failure if they responded otherwise.
Time Frame: Outcome was measured at three months following randomization.
Population: If participant did not attend the three-month follow-up, missing values were imputed by either the value from the next available follow-up or if the participant was lost to follow-up the participant was treated as a failure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pessary | Behavioral Therapy | Combination of Pessary and Behavioral Therapy
Number analyzed (Participants) | 149 | 146 | 150
Participants | 80 | 72 | 59
Statistical Analysis 1: Comparison: Pessary vs Behavioral Therapy; A priori, the combination treatment was considered superior (75% success rate) to either single-modality therapy (60% success rate) at 80% power with 150 participants per group; Test type: Non-Inferiority — Logistic regression was used to adjust for randomization stratification variables of incontinence type and incontinence severity. No parameter estimates were reported. No adjustments for multiple comparisons made; p < 0.0492, Regression, Logistic — A priori threshold for statistical significance set at p = 0.0492 to account for interim analysis
Statistical Analysis 2: Comparison: Pessary vs Combination of Pessary and Behavioral Therapy; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.02, Regression, Logistic — A priori threshold for statistical significance set at p = 0.0492 to account for interim analysis
Statistical Analysis 3: Comparison: Behavioral Therapy vs Combination of Pessary and Behavioral Therapy; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.49, Regression, Logistic — A priori threshold for statistical significance set at p = 0.0492 to account for interim analysis

2. Primary Outcome: No Bothersome Stress Incontinence Symptoms at 3 Months
Description: Success if participants answer either "no" or "yes" with a bother component of "not at all" or "somewhat" to all seven Urogenital Distress Inventory-Stress Incontinence Subscale items of the Pelvic Floor Distress Inventory, or a failure if they responded otherwise.
Time Frame: Outcome was measured at three months following randomization.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pessary | Behavioral Therapy | Combination of Pessary and Behavioral Therapy
Number analyzed (Participants) | 149 | 146 | 150
Participants | 66 | 71 | 49
Statistical Analysis 1: Comparison: Pessary vs Behavioral Therapy; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.006, Regression, Logistic
Statistical Analysis 2: Comparison: Pessary vs Combination of Pessary and Behavioral Therapy; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.048, Regression, Logistic
Statistical Analysis 3: Comparison: Behavioral Therapy vs Combination of Pessary and Behavioral Therapy; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.42, Regression, Logistic

3. Secondary Outcome: "Much Better" or "Very Much Better" on PGI-I at 12 Months
Description: as for outcome 1
Time Frame: Outcome was measured at 12 months following randomization.
Population: If participant did not attend the 12-month follow-up, missing values were imputed as a failure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pessary | Behavioral Therapy | Combination of Pessary and Behavioral Therapy
Number analyzed (Participants) | 149 | 146 | 150
Participants | 49 | 48 | 47
Statistical Analysis 1: Comparison: Pessary vs Behavioral Therapy; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0492, Regression, Logistic
Statistical Analysis 2: Comparison: Pessary vs Combination of Pessary and Behavioral Therapy; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0492, Regression, Logistic
Statistical Analysis 3: Comparison: Behavioral Therapy vs Combination of Pessary and Behavioral Therapy; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0492, Regression, Logistic

4. Secondary Outcome: No Bothersome Stress Incontinence Symptoms at 12 Months.
Description: as for outcome 2
Time Frame: Outcome was measured at 12 months following randomization.
Population: If participant did not attend the 12-month follow-up, missing values were imputed as a failure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pessary | Behavioral Therapy | Combination of Pessary and Behavioral Therapy
Number analyzed (Participants) | 149 | 146 | 150
Participants | 49 | 59 | 52
Statistical Analysis 1: Comparison: Pessary vs Behavioral Therapy; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0492, Regression, Logistic
Statistical Analysis 2: Comparison: Pessary vs Combination of Pessary and Behavioral Therapy; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0492, Regression, Logistic
Statistical Analysis 3: Comparison: Behavioral Therapy vs Combination of Pessary and Behavioral Therapy; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0492, Regression, Logistic

5. Secondary Outcome: 75% Reduction in Weekly Urinary Incontinence Episodes at 3 Months
Description: Success if participants reported at least 75% reduction in frequency of incontinence episodes on 7-day bladder diary, a failure if they reported otherwise.
Time Frame: Outcome was measured at three months following randomization.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pessary | Behavioral Therapy | Combination of Pessary and Behavioral Therapy
Number analyzed (Participants) | 149 | 146 | 150
Participants | 80 | 68 | 69
Statistical Analysis 1: Comparison: Pessary vs Behavioral Therapy; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0492, Regression, Logistic
Statistical Analysis 2: Comparison: Pessary vs Combination of Pessary and Behavioral Therapy; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0492, Regression, Logistic
Statistical Analysis 3: Comparison: Behavioral Therapy vs Combination of Pessary and Behavioral Therapy; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0492, Regression, Logistic

6. Secondary Outcome: 75% Reduction in Weekly Urinary Incontinence Episodes at 12 Months
Description: as for outcome 5
Time Frame: Outcome was measured at 12 months following randomization.
Population: If participant did not attend the 12-month follow-up, missing values were imputed as a failure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pessary | Behavioral Therapy | Combination of Pessary and Behavioral Therapy
Number analyzed (Participants) | 149 | 146 | 150
Participants | 52 | 54 | 51
Statistical Analysis 1: Comparison: Pessary vs Behavioral Therapy; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0492, Regression, Logistic
Statistical Analysis 2: Comparison: Pessary vs Combination of Pessary and Behavioral Therapy; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0492, Regression, Logistic
Statistical Analysis 3: Comparison: Behavioral Therapy vs Combination of Pessary and Behavioral Therapy; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0492, Regression, Logistic

7. Secondary Outcome: Satisfaction With Treatment at 3 Months
Description: Success if participant reported being "satisfied" on Patient Satisfaction Question (PSQ), a failure if they reported otherwise.
Time Frame: Outcome was measured at three months following randomization.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pessary | Behavioral Therapy | Combination of Pessary and Behavioral Therapy
Number analyzed (Participants) | 149 | 146 | 150
Participants | 118 | 110 | 94
Statistical Analysis 1: Comparison: Pessary vs Behavioral Therapy; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.03, Regression, Logistic
Statistical Analysis 2: Comparison: Pessary vs Combination of Pessary and Behavioral Therapy; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.048, Regression, Logistic
Statistical Analysis 3: Comparison: Behavioral Therapy vs Combination of Pessary and Behavioral Therapy; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0492, Regression, Logistic

8. Secondary Outcome: Satisfaction With Treatment at 12 Months
Description: as for outcome 7
Time Frame: Outcome was measured at 12 months following randomization.
Population: If participant did not attend the 12-month follow-up, missing values were imputed as a failure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pessary | Behavioral Therapy | Combination of Pessary and Behavioral Therapy
Number analyzed (Participants) | 149 | 146 | 150
Participants | 81 | 79 | 75
Statistical Analysis 1: Comparison: Pessary vs Behavioral Therapy; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0492, Regression, Logistic
Statistical Analysis 2: Comparison: Pessary vs Combination of Pessary and Behavioral Therapy; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0492, Regression, Logistic
Statistical Analysis 3: Comparison: Behavioral Therapy vs Combination of Pessary and Behavioral Therapy; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0492, Regression, Logistic

ADVERSE EVENTS:
Time Frame: Adverse events were collected during treatment visits over an 8-week treatment period.
Description: As no other adverse events, those that don't meet the definition of a SAE, occurred in at least 5% of participants in any one of the three arms for the ATLAS trial, no table was generated as it is not required by law.
Arm/Group | Pessary | Behavioral Therapy | Combination of Pessary and Behavioral Therapy
Serious Adverse Events (participants affected / at risk) | 7/149 | 4/146 | 6/150
Other Adverse Events (participants affected / at risk) | 0/149 | 0/146 | 0/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pessary (N=149) | Behavioral Therapy (N=146) | Combination of Pessary and Behavioral Therapy (N=150)
Urinary incontinence surgery (Renal and urinary disorders) | 2 (2) | 0 (0) | 2 (2)
Cholecystectomy (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Angioplasty of heart (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hiatal hernia repair (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Left femoral hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Left eye surgery for cancer (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain and anxiety (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Oophorectomy (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fractured right leg and ankle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lumbar decompression surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Right knee surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Kidney surgery (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Uterine cancer (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No